CLINICAL TRIAL: NCT04451317
Title: Changes in Physical and Sports Activity, Anxiety and Sleep Patterns Following the Containment Period Imposed by the COVID-19 Pandemic in Patients With Chronic Medical Conditions and in Healthy Athletes.
Brief Title: Physical Activity Following the Containment Period Imposed by the COVID-19 Pandemic in Patients
Acronym: PhysiCOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0203
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Physical Activity; COVID-19
Keywords: anxiety; sleep; chronic pathology
MeSH Terms: conditions — Motor Activity; COVID-19; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Patients involved in a Sport-Health initiative Visit once by telephone and then ask to fill in 3 questionnaires on a digital platform within 48 hours after the telephone interview.
  Interventions: Other: Questionnaire, phone call
- Control: Healthy sport subjects. Visit once by telephone and then ask to fill in 3 questionnaires on a digital platform within 48 hours after the telephone interview.
  Interventions: Other: Questionnaire, phone call

INTERVENTIONS:
Other: Questionnaire, phone call — phone call and 3 questionnaires on a digital platform

SUMMARY:
In the context of the containment imposed by the COVID-19 pandemic and taking into account the numerous restrictions imposed, the practice of physical and sports activities (PSA) could be reduced by general population and sports population. While the practice of regular physical activity (PA) is prescribed and widely recognized as effective for the management of many chronic conditions and that regular participation in sports (SA) reduces the risk of injury and cardiac accidents- vascular disease in sports subjects, the reduction in regular physical activity levels in the wake of the period of confinement is likely to induce a medical risk in connection with the resumption of PSA.

DETAILED DESCRIPTION:
The study is non-interventional. The data that will be collected are data that can be integrated into a care procedure in accordance with the recommendations to accompany the patients with chronic pathology and athletes for the resumption of PSA after hypothetical deconditioning. Support will be implemented in accordance with the recommendations of the HCSP and the Ministry of Sports. The objective of this study is to evaluate the data of this recommended medical follow-up.

The questionnaires used for the subjects' self-evaluation are all validated in French language, used in the context of medical monitoring, and used in clinical research: assessment of physical activity levels by the questionnaire of RICCI and GAGNON (RG), evaluation of the level of Anxiety and Depression by the Hospital and Anxiety Scale Depression (AHH), assessment of sleep quality by the score of LEEDS.

Medical questionnaires to assess the evolutionary stage of chronic pathologies (MS, Parkinson's disease and Fibromyalgia) will be informed by the investigating physician during the interview telephone with the patient.

ELIGIBILITY:
Inclusion Criteria:

* non-working or tele-working subjects, subjects who have returned to work, subjects who have taken up a part-time professional activity, subjects who have resumed an activity full-time professional
* subjects who have given their consent
* for the sports topics group: amateur level (no sportsmen and women professionals), including sports subjects in the disabled category, with no chronic pathology, already followed by the investigating medical units.
* for the group of patients with chronic diseases: subjects carrying a chronic pathology (rheumatic pathologies, etc) and fibromyalgia, Parkinson's disease and multiple sclerosis, cancer of the breast, metabolic diseases without cardiovascular failure) usually accompanied by the medical units for the implementation of a programme of physic adapted and medically prescribed (Sport-Santé approach)
* social security affiliation

Exclusion Criteria:

* Patient under the protection of adults (guardianship, curators), safeguard of justice),
* Pregnant and/or breastfeeding woman.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: healthy athletes or patients involved in a Sport-health initiative
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Physical activity measure | 1 day
  Changes in the level of physical activity (questionnaire from RICCI-GAGNON)

SECONDARY OUTCOMES:
Depression | 1 day
  To evaluate the f the level of anxiety and depression by questionnaire HAD
Sleep quality | 1 day
  To evaluate the level of sleep activity by questionnaire LEEDS
food activity | 1 day
  To evaluate the food activity by questionnaire LEEDS
activity level of chronic pathology | 1 day
  To evaluate of the activity level of chronic pathology (monitoring criteria in accordance with good clinical practice) in patients with chronic pathology by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Pillard, MD, Principal Investigator — University Hopsital Toulouse
Locations (2):
- France (2):
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse